CLINICAL TRIAL: NCT05403411
Title: The Effect of Two Different Education Methods Based on Distance Education for Nursing Students on Critical Thinking
Brief Title: Distance Education for Nursing Students on Critical Thinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Tayaz (Other)
Responsible Party: Sponsor-Investigator, Esra Tayaz, Research Assistant, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-127
Record Dates: First submitted 2022-05-22; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Critical Thinking
Keywords: Critical thinking; Intensive care; Nursing student; Distance education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Distance education for nursing students on critical thinking
  Interventions: Other: Distance education for nursing students on critical thinking
- Control group (No Intervention): The control group was given a booklet for critical thinking.

INTERVENTIONS:
Other: Distance education for nursing students on critical thinking — The students in the intervention group were trained with distance education method for the first 4 weeks, and in the following weeks, with theoretical and case presentations. Critical thinking techniques were used during the trainings. A total of 8 weeks of training was given. Training was given for the first 5 weeks without interruption, and for the next three weeks with a two-week break. Critical thinking disposition scale was applied in the pre-test and post-test.
  Arms: Intervention group

SUMMARY:
Critical thinking forms the basis of nursing knowledge. Critical thinking skills constitute a vital part of the nurse's work performance, adaptation, problem solving, awareness of the responsibilities of the profession, and the conceptual understanding of nursing. Due to the increasing number of dependent patients, complex care needs and increasing research in the field of health, intensive care nurses have to think critically in order to learn throughout life, develop professionally, work effectively with teammates, reach care and treatment goals, and contribute to the change of society.

DETAILED DESCRIPTION:
The sample size of the study was calculated using the G*Power Software (ver. 3.1.9.2) program. For the smallest sample size of the study, 85% power and medium effect size (f:0.25) at the 95% confidence interval, 110 individuals were found, with at least 55 individuals in each group. The intervention group consisted of students enrolled in the intensive care nursing course, which is one of the third year elective courses, and the control group consisted of the students enrolled in the perinatology course from the third year elective courses. The study was completed on a voluntary basis. After the losses, a sample of 64 from the intervention group and 54 from the control group was created, and the data of a total of 118 students were evaluated. The students in the intervention group were given theoretical training for the first 4 weeks, followed by theoretical and case presentations in the following weeks. It is aimed to increase the critical thinking disposition of the students by using critical thinking techniques during the trainings. A total of 8 weeks of training was given. For the first 5 weeks, training was given with a two-week break for the next three weeks. The control group was given a booklet for critical thinking. Pre-test and post-test were applied simultaneously to both groups. Critical thinking disposition scale was applied in the pre-test and post-test.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the research,
* Willingness to participate in the research,
* Not having taken a critical thinking course before,
* Being able to speak Turkish,

Exclusion Criteria:

* Not being willing to participate in the research,
* Not willing to participate in the research,
* To fill in the research forms incompletely,
* Working as a nurse in an institution
* To be a graduate of the nursing department from a health vocational high school.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
critical thinking disposition | before the implementation
  evaluated with "critical thinking disposition (CTHD) scale". This scale include 5 subdimensions. Total minimum score is 49, maximum score is 245. An increase in the score indicates that the tendency to think critically increases.
critical thinking disposition | 8 weeks after the implementation
  evaluated with "critical thinking disposition (CTHD) scale". This scale include 5 subdimensions. Total minimum score is 49, maximum score is 245. An increase in the score indicates that the tendency to think critically increases.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tayaz, Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No